CLINICAL TRIAL: NCT07198438
Title: A Block-Randomized Study Comparing Deep and Standard Prolonged Intermittent Theta Burst Stimulation on Emotional Symptoms and Physiological Indicators in Patients With Major Depression
Brief Title: Deep Versus Standard Prolonged Intermittent Theta Burst Stimulation for Depression
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202506034RINB
Record Dates: First submitted 2025-09-21; First posted 2025-09-30 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Intermittent Theta Burst Stimulation; Repetitive Transcranial Magnetic Stimulation; Depression
Keywords: Repetitive Transcranial Magnetic Stimulation; intermittent theta burst stimulation; depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The raters for the primary and key secondary outcome scales (including HAM-D17, HAM-A, YMRS, and Y-BOCS) are blinded to the participant's treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep piTBS (Experimental): Participants assigned to the experimental group receive prolonged intermittent theta burst stimulation (piTBS) with a double-cone coil targeting the anterior cingulate cortex (ACC).
  Interventions: Device: Deep Prolonged Intermittent Theta Burst Stimulation
- Standard piTBS (Active Comparator): Participants assigned to the active comparator group receive prolonged intermittent theta burst stimulation (piTBS) with a planar coil targeting the left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Standard Prolonged Intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: Deep Prolonged Intermittent Theta Burst Stimulation — This intervention uses a Deymed Repetitive Transcranial Magnetic Stimulator with a double-cone coil (90BFVT-LQC) to target the anterior cingulate cortex (ACC). The resting motor threshold (rMT) is determined from the tibialis anterior muscle. Stimulation is delivered at 90% of the rMT. The protocol consists of 3-pulse 50Hz bursts repeated at a 5Hz frequency, administered in cycles of 2 seconds on and 8 seconds off, for a total of 1800 pulses per session. Treatment consists of 20 sessions administered over four weeks.
  Arms: Deep piTBS
Device: Standard Prolonged Intermittent Theta Burst Stimulation — This intervention uses a Deymed Repetitive Transcranial Magnetic Stimulator with a planar coil (70BF-LQC) to target the left dorsolateral prefrontal cortex (DLPFC). The resting motor threshold (rMT) is determined from the abductor pollicis brevis muscle. The DLPFC is localized using Beam F3 method. Stimulation is delivered at 90% of the rMT. The protocol consists of 3-pulse 50Hz bursts repeated at a 5Hz frequency, administered in cycles of 2 seconds on and 8 seconds off, for a total of 1800 pulses per session. Treatment consists of 20 sessions administered over four weeks.
  Arms: Standard piTBS

SUMMARY:
This study compares two types of non-invasive brain stimulation to treat major depression in patients who have not found relief from at least one antidepressant medication.

The study will use a specific type of brain stimulation called prolonged intermittent Theta Burst Stimulation (piTBS). The standard way to use piTBS for depression is to target an area on the side of the head called the dorsolateral prefrontal cortex (DLPFC). This study will compare this standard piTBS method with a newer approach, deep piTBS, which targets a different, deeper area in the middle of the brain called the anterior cingulate cortex (ACC).

Participants will be randomly assigned to one of two groups. One group will receive the deep piTBS treatment, and the other will receive the standard piTBS treatment. Both treatments are given once a day, five days a week, for four weeks. The study aims to find out if the deep piTBS approach is more effective at reducing symptoms of depression than the standard approach. Researchers will also look at effects on anxiety and other related symptoms.

DETAILED DESCRIPTION:
Background:

Major depressive disorder (MDD) is associated with dysfunction in large-scale brain networks, including the central executive network (CEN), default mode network (DMN), and the salience network (SN). The anterior cingulate cortex (ACC) is a key hub in the SN, and its dysfunction is believed to be a core pathological feature of depression. While high-frequency repetitive transcranial magnetic stimulation (rTMS) over the left dorsolateral prefrontal cortex (DLPFC) is an evidence-based treatment for treatment-resistant depression (TRD), it only indirectly modulates deeper structures like the ACC. Deep TMS techniques using a double-cone coil can directly stimulate deeper regions such as the medial prefrontal cortex (mPFC) and ACC, which may offer a more direct and potentially more effective therapeutic approach. Intermittent theta burst stimulation (iTBS) is a newer form of rTMS that significantly shortens treatment time, but its application to deep brain targets like the ACC has not been well-studied.

Objective:

This study aims to compare the therapeutic efficacy of prolonged intermittent theta burst stimulation (piTBS) targeting the ACC (deep piTBS) versus the standard protocol targeting the left DLPFC (standard piTBS) for patients with TRD. The study will also evaluate the effects of these interventions on comorbid anxiety, obsessive-compulsive, and somatic symptoms, as well as on physiological indicators.

Study Design:

This is a single-center, block-randomized study. A maximum of 90 participants meeting DSM-5 criteria for major depressive disorder, who have failed to respond to at least one adequate trial of an antidepressant, will be recruited. Participants will be randomly assigned in a 2:1 ratio (deep piTBS: standard piTBS, within blocks of six) to one of two treatment arms:

Deep piTBS Group: Participants will receive stimulation targeting the ACC using a double-cone coil. Stimulation intensity will be set at 90% of the resting motor threshold (rMT) determined from the tibialis anterior muscle.

Standard piTBS Group: Participants will receive stimulation targeting the left DLPFC using a standard figure-8 coil. Intensity will be set at 90% of the rMT determined from the abductor pollicis brevis muscle.

For both groups, the piTBS protocol consists of 1800 pulses per session, delivered daily (5 days/week) for 4 weeks, for a total of 20 sessions.

Outcome Measures:

The primary outcome is the change in the 17-item Hamilton Depression Rating Scale (HAM-D17) score from baseline to the end of treatment (after 20 sessions). Secondary outcomes include changes in scores on the Hamilton Anxiety Rating Scale (HAM-A), Yale-Brown Obsessive Compulsive Scale (Y-BOCS), Patient Health Questionnaire-15 (PHQ-15), Beck Depression Inventory-II (BDI-II), Beck Anxiety Inventory (BAI), and various physiological measures including heart rate variability (HRV). Assessments will be conducted at baseline, after every 5 treatment sessions, and one week after the completion of the 20th session.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 70 years, inclusive.
* Diagnosis of Major Depressive Disorder (MDD) with a current major depressive episode, according to DSM-5 criteria, as confirmed by a psychiatrist.
* History of inadequate response to at least one trial of an antidepressant medication of adequate dose and duration.
* A score of 18 or greater on the 17-item Hamilton Depression Rating Scale (HAM-D17) at the screening visit.

Exclusion Criteria:

* Lifetime diagnosis of any primary psychotic disorder (e.g., schizophrenia spectrum disorders) or bipolar and related disorders according to DSM-5.
* Significant current suicide risk, as indicated by a score of 4 on item 3 of the HAM-D17.
* Current substance use disorder (excluding tobacco) within the last 3 months, according to DSM-5.
* Presence of significant cognitive impairment, such as intellectual disability, delirium, or a diagnosed neurocognitive disorder.
* Any personal history of seizures, stroke, brain tumor, brain aneurysm, increased intracranial pressure, or other major neurological disorders.
* Presence of metal implants in the head (excluding dental fillings) or any implanted medical devices such as a cardiac pacemaker or defibrillator.
* Currently pregnant.
* Any other major medical condition that, in the investigator's judgment, could compromise participant safety or interfere with the study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the 17-item Hamilton Depression Rating Scale (HAM-D17) Score | Baseline (Day 1, prior to first treatment), after 5 treatments (Week 1), after 10 treatments (Week 2), after 15 treatments (Week 3), after 20 treatments (End of Week 4), and at a 1-week follow-up after the final treatment session.
  The 17-item Hamilton Depression Rating Scale (HAM-D17) is a clinician-rated scale that assesses the severity of depressive symptoms. The total score is derived from a structured interview conducted by a trained outcomes assessor who is blinded to the participant's treatment group. Scores range from 0-52, where higher scores indicate more severe depression.

SECONDARY OUTCOMES:
Change From Baseline in the Hamilton Anxiety Rating Scale (HAM-A) Score | Baseline (prior to first treatment), after 5 treatments (Week 1), after 10 treatments (Week 2), after 15 treatments (Week 3), after 20 treatments (End of Week 4), and at a 1-week follow-up after the final treatment session.
  The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-rated scale used to assess the severity of anxiety symptoms. A trained outcomes assessor, who is blinded to the participant's treatment group, determines the score based on a clinical interview. Higher scores indicate more severe anxiety.
Change From Baseline in the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) Score | Baseline (prior to first treatment), after 5 treatments (Week 1), after 10 treatments (Week 2), after 15 treatments (Week 3), after 20 treatments (End of Week 4), and at a 1-week follow-up after the final treatment session.
  The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is a clinician-rated scale designed to measure the severity of obsessive-compulsive symptoms. The score is determined through an interview conducted by a trained outcomes assessor who is blinded to the treatment allocation. Higher scores reflect greater symptom severity.
Change From Baseline in the Beck Depression Inventory-II (BDI-II) Score | Baseline (prior to first treatment), after 5 treatments (Week 1), after 10 treatments (Week 2), after 15 treatments (Week 3), after 20 treatments (End of Week 4), and at a 1-week follow-up after the final treatment session.
  The Beck Depression Inventory-II (BDI-II) is a 21-item self-report questionnaire designed to measure the severity of depression. Participants rate various depressive symptoms based on their experiences over the past two weeks. This scale provides a patient-reported perspective on depression, complementing the clinician-rated HAM-D17. Higher scores indicate greater depression severity.
Change From Baseline in the Beck Anxiety Inventory (BAI) Score | Baseline (prior to first treatment), after 5 treatments (Week 1), after 10 treatments (Week 2), after 15 treatments (Week 3), after 20 treatments (End of Week 4), and at a 1-week follow-up after the final treatment session.
  The Beck Anxiety Inventory (BAI) is a 21-item self-report scale that measures the severity of anxiety symptoms. It is completed by the participant and assesses how much they have been bothered by common symptoms of anxiety over the past week. This serves as a patient-reported measure of anxiety, complementing the clinician-rated HAM-A. Higher scores indicate greater anxiety levels.
Change From Baseline in the Young Mania Rating Scale (YMRS) Score | Baseline (prior to first treatment), after 5 treatments (Week 1), after 10 treatments (Week 2), after 15 treatments (Week 3), after 20 treatments (End of Week 4), and at a 1-week follow-up after the final treatment session.
  The Young Mania Rating Scale (YMRS) is an 11-item, clinician-rated scale used to evaluate the severity of manic symptoms. It is administered via interview by a trained assessor who is blinded to the treatment group. In this study, it is used to monitor for potential treatment-emergent mania or hypomania. Higher scores indicate more severe manic symptoms.
Change From Baseline in the Patient Health Questionnaire-15 (PHQ-15) Score | Baseline (prior to first treatment), after 5 treatments (Week 1), after 10 treatments (Week 2), after 15 treatments (Week 3), after 20 treatments (End of Week 4), and at a 1-week follow-up after the final treatment session.
  The Patient Health Questionnaire-15 (PHQ-15) is a self-report scale that assesses the severity of 15 common somatic symptoms. This questionnaire is completed by the participant. Higher scores indicate greater somatic symptom severity.
Change From Baseline in the Health Anxiety Questionnaire (HAQ) Score | Baseline (prior to first treatment), after 5 treatments (Week 1), after 10 treatments (Week 2), after 15 treatments (Week 3), after 20 treatments (End of Week 4), and at a 1-week follow-up after the final treatment session.
  The Health Anxiety Questionnaire (HAQ) is a self-report scale designed to measure the severity of health-related anxiety. Participants rate their health-related worries and beliefs. Higher scores indicate a greater degree of health anxiety. It is a self-administered questionnaire.
Change From Baseline in Heart Rate Variability (HRV) Indices | Baseline (prior to first treatment), after 5 treatments (Week 1), after 10 treatments (Week 2), after 15 treatments (Week 3), after 20 treatments (End of Week 4), and at a 1-week follow-up after the final treatment session.
  Heart Rate Variability (HRV) is a physiological measure of autonomic nervous system function, measured using an electrocardiogram (EKG). Specific indices will be analyzed, including the ratio of low-frequency to high-frequency power (LF/HF) and the standard deviation of normal to normal RR intervals (SDNN).
Change From Baseline in Skin Conductance | Baseline (prior to first treatment), after 5 treatments (Week 1), after 10 treatments (Week 2), after 15 treatments (Week 3), after 20 treatments (End of Week 4), and at a 1-week follow-up after the final treatment session.
  Skin conductance is a physiological measure of electrodermal activity that reflects sympathetic nervous system arousal. It is measured non-invasively via electrodes placed on the skin to assess changes in physiological arousal levels throughout the course of treatment.
Change From Baseline in Respiratory Sinus Arrhythmia (RSA) | Baseline (prior to first treatment), after 5 treatments (Week 1), after 10 treatments (Week 2), after 15 treatments (Week 3), after 20 treatments (End of Week 4), and at a 1-week follow-up after the final treatment session.
  Respiratory Sinus Arrhythmia (RSA) is the naturally occurring variation in heart rate that occurs during the breathing cycle. It is considered a key measure of parasympathetic nervous system activity (vagal tone) and is derived from simultaneously recorded electrocardiogram (EKG) and respiratory signals.
Change From Baseline in Finger Temperature | Baseline (prior to first treatment), after 5 treatments (Week 1), after 10 treatments (Week 2), after 15 treatments (Week 3), after 20 treatments (End of Week 4), and at a 1-week follow-up after the final treatment session.
  Finger temperature is a physiological measure of peripheral blood flow, which is influenced by the autonomic nervous system. It is measured non-invasively and used as an indicator of physiological stress and arousal.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hao Ma, MD, Principal Investigator — Department of Psychiatry, National Taiwan University Hospital, Yunlin Branch
Locations (1):
- Department of Psychiatry, National Taiwan University Hospital, Yunlin Branch, Douliu, Yunlin County, Taiwan

IPD SHARING:
Plan to Share IPD: No